CLINICAL TRIAL: NCT06899958
Title: Metabolism Enhancement by Laser Therapy
Acronym: MELT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maria Alora, Director, MGH Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000547
Record Dates: First submitted 2025-03-18; First posted 2025-03-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metabolism Disorder
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fractional Laser treatment (Experimental): Large Area Fractional Laser treatments to the abdomen and thighs using the MIRIA laser.
  Interventions: Device: Fractional Laser

INTERVENTIONS:
Device: Fractional Laser — Three fractional laser treatments to the abdomen and thighs at 4 week intervals.

SUMMARY:
This is a single-center, open-label pilot study to determine the effect of large area fractional laser treatment (LAFLT) on adults' metabolic profile.

DETAILED DESCRIPTION:
The current research project aims to investigate the effects of large-area fractional laser treatment (LAFLT) on body weight, metabolism, and body composition. Prior research suggests that treating large skin areas with fractional laser therapy may stimulate metabolism and promote weight loss. The MIRIA laser, an FDA-approved fractional laser, is widely used for skin aging, acne scarring, and wrinkle reduction and will be used to evaluate these potential metabolic effects.

Subjects aged 18-60 with a BMI of 25-30 will undergo three fractional laser treatments on the abdomen and thighs over 36 weeks, with sessions every four weeks. The study includes six total visits, incorporating photography, non-invasive imaging, x-rays, blood draws, and two optional biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. 18- 60 years of age;
2. BMI between 25.0 and 30 kg/m2;
3. Subjects must be in good general health, based on answers provided during the screening visit;
4. Subject must be able and willing to provide written informed consent and comply with the requirements of the study protocol.
5. Females of childbearing potential must be willing and able to use a medically highly effective form of birth control during the entire study.

Exclusion Criteria:

1. Participation in another investigational drug or device clinical trial in the past 30 days;
2. Currently pregnant or pregnancy within the past 6 months or currently breastfeeding;
3. Have a history of drug or alcohol abuse in the past 3 years or have reported habitual alcohol intake greater than 2 standard drinks per day (e.g., 2 beers, 2 glasses of wine, or 2 mixed drinks);
4. Planning or currently participating in a weight loss program;
5. Plan to change daily diet or level of physical activity;
6. Intake of medication that may affect body weight such as GLP-1 receptor agonists, amitriptyline, bupropion, thyroid medications, etc.;
7. History of cancer which required lymph node biopsy or dissection;
8. Weight loss or gain of 10 kg or more in the past 6 months;
9. History of diabetes mellitus or cardiac disease;
10. Intake of hormone replacement therapy (HRT) in the last 6 months;
11. Infection, surgery, or history of trauma or laser treatment to the treatment area in the past 6 months;
12. Presence of any skin disease on the abdomen or thighs;
13. Have birthmarks, tattoos, scars, or any other disfiguration of the skin in the abdomen or thighs;
14. Presence of sunburn or tan in the abdomen or thighs;
15. Use of any topical application of retinoids in the past 6 weeks on the abdomen or thighs or intake of systemic retinoids in the past 6 months;
16. Use of any prescription topical medication, such as corticosteroids or hydroquinone on the abdomen or thighs in the past 6 weeks;
17. History of keloid formation or hypertrophic scarring;
18. History of bariatric surgery or other major weight-loss procedures;
19. History of abdominal liposuction, abdominoplasty or CoolSculpting;
20. Known allergy to lidocaine or other local anesthetics;
21. The investigator believes that the subject is an unsuitable candidate to participate in the study, receive laser treatment, or would be placed at risk by participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Body Fat (%) | Week 1, 12, 24
  The percent body fat will be collected from the Dual energy x-ray absorptiometry scan (DEXA) and via the Bioelectrical Impedance Analysis (BIA).
Body Mass Index (BMI) (kg/m²) | Week 0, 4, 8, 12, 24
  BMI will be calculated using the formula: weight (kg) / [height (m)]². Height will be measured at the baseline visit and body weight will be measured at each of the following visits.
Waist circumference (cm) | Week 0, 4, 8, 12, 24
  These measurements will be taken at each of the following visits
Hip circumference (cm) | Week 0, 4, 8, 12, 24
  These measurements will be taken at each of the following visits
Arm circumference (cm) | Week 0, 4, 8, 12, 24
  These measurements will be taken at each of the following visits
Total Lean Body Mass (kg) | Week 1, 12, 24
  The total lean body mass will be collected from the Dual energy x-ray absorptiometry scan (DEXA) and via the Bioelectrical Impedance Analysis (BIA).

SECONDARY OUTCOMES:
Complete Blood Count (CBC) | Week 0, 4, 8, 12, 24
  Measurement of red blood cell count, white blood cell count, hemoglobin, hematocrit, and platelet count via a blood draw.
Comprehensive Metabolic Panel (CMP) | Week 0, 4, 8, 12, 24
  Assessment of glucose, calcium, electrolyte and fluid balance (sodium, potassium, CO2, chloride), kidney function (BUN, creatinine), and liver function (albumin, total protein, ALP, ALT, AST, bilirubin) via a blood draw.
Lipid Panel | Week 0, 4, 8, 12, 24
  Measurement of total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides via a blood draw.
HbA1c | Week 0, 4, 8, 12, 24
  Measurement of hemoglobin A1c via a blood draw.
C-Reactive Protein (CRP) | Week 0, 4, 8, 12, 24
  Measurement of CRP levels via a blood draw.
Erythrocyte Sedimentation Rate (ESR) | Week 0, 4, 8, 12, 24
  Assessment of the rate at which red blood cells sediment via a blood draw.
Histamine | Week 0, 4, 8, 12, 24
  Measurement of plasma histamine levels via a blood draw.
Cortisol | Week 0, 4, 8, 12, 24
  Measurement of serum cortisol levels via a blood draw.
Oxytocin | Week 0, 4, 8, 12, 24
  Measurement of serum oxytocin levels via a blood draw.
Creatine Phosphokinase (CPK) | Week 0, 4, 8, 12, 24
  Measurement of serum CPK via a blood draw.
Serum Interleukin-6 (IL-6) | Week 0, 4, 8, 12, 24
  Measurement of interleukin-6 (IL-6) via a blood draw.
Serum Norepinephrine | Week 0, 4, 8, 12, 24
  Measurement of norepinephrine via a blood draw.
Indirect Calorimetry | Week 0,12, 24
  This is a non-invasive procedure that measures how much energy the body uses.
Skin Biopsy (Optional) | Week 1, 12
  2 optional biopsies will be take pre- and post-laser treatment to measure changes in collagen and skin thickness.
Skin Elasticity | Week 0, 4, 8, 12, 24
  Ultrasound will be used to measure skin elasticity.
Skin Thickness | Week 0, 4, 8, 12, 24
  Ultrasound will be used to measure skin thickness.
Hydration Status (%) | Week 0, 12
  Estimation of total body water content as a percentage of body weight using the Bioelectrical impedance analysis (BIA).
VAS Pain Score | Week 1, 4, 8
  The visual analog scale (VAS) pain score will be collected from the subject after each laser treatment. The VAS is a 10cm long scale with 0cm representing "no pain" and 10cm representing "worst possible pain".
Total Body Bone Mineral Density (g/cm²) | Week 1, 12, 24
  The total body BMD will be collected from the Dual energy x-ray absorptiometry scan (DEXA).

CONTACTS AND LOCATIONS:
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Salma N, Wang-Evers M, Karasik D, Yerevanian A, Downs H, Luo T, Doyle AE, Tannous Z, Cacicedo JM, Manstein D. Large area fractional laser treatment of mouse skin increases energy expenditure. iScience. 2023 Dec 7;27(1):108677. doi: 10.1016/j.isci.2023.108677. eCollection 2024 Jan 19. PMID 38213618
- [Background] May M, Schindler C, Engeli S. Modern pharmacological treatment of obese patients. Ther Adv Endocrinol Metab. 2020 Jan 22;11:2042018819897527. doi: 10.1177/2042018819897527. eCollection 2020. PMID 32030121
- [Background] Singh G, Krauthamer M, Bjalme-Evans M. Wegovy (semaglutide): a new weight loss drug for chronic weight management. J Investig Med. 2022 Jan;70(1):5-13. doi: 10.1136/jim-2021-001952. Epub 2021 Oct 27. PMID 34706925
- [Background] Bettini S, Belligoli A, Fabris R, Busetto L. Diet approach before and after bariatric surgery. Rev Endocr Metab Disord. 2020 Sep;21(3):297-306. doi: 10.1007/s11154-020-09571-8. PMID 32734395
- [Background] Patsouris D, Qi P, Abdullahi A, Stanojcic M, Chen P, Parousis A, Amini-Nik S, Jeschke MG. Burn Induces Browning of the Subcutaneous White Adipose Tissue in Mice and Humans. Cell Rep. 2015 Nov 24;13(8):1538-44. doi: 10.1016/j.celrep.2015.10.028. Epub 2015 Nov 12. PMID 26586436
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Laubach HJ, Tannous Z, Anderson RR, Manstein D. Skin responses to fractional photothermolysis. Lasers Surg Med. 2006 Feb;38(2):142-9. doi: 10.1002/lsm.20254. PMID 16392146
- [Background] Gotkin RH, Sarnoff DS, Cannarozzo G, Sadick NS, Alexiades-Armenakas M. Ablative skin resurfacing with a novel microablative CO2 laser. J Drugs Dermatol. 2009 Feb;8(2):138-44. PMID 19213229
- [Background] Prignano F, Ricceri F, Bonan P, Cannarozzo G, Campolmi P. Induction of apoptosis by fractional CO2 laser treatment. J Cosmet Laser Ther. 2012 Dec;14(6):267-71. doi: 10.3109/14764172.2012.738820. PMID 23058108
- [Background] Bogdan Allemann I, Kaufman J. Fractional photothermolysis--an update. Lasers Med Sci. 2010 Jan;25(1):137-44. doi: 10.1007/s10103-009-0734-8. PMID 19787413
- [Background] Porter C, Tompkins RG, Finnerty CC, Sidossis LS, Suman OE, Herndon DN. The metabolic stress response to burn trauma: current understanding and therapies. Lancet. 2016 Oct 1;388(10052):1417-1426. doi: 10.1016/S0140-6736(16)31469-6. PMID 27707498
- [Background] Knuth CM, Auger C, Jeschke MG. Burn-induced hypermetabolism and skeletal muscle dysfunction. Am J Physiol Cell Physiol. 2021 Jul 1;321(1):C58-C71. doi: 10.1152/ajpcell.00106.2021. Epub 2021 Apr 28. PMID 33909503
- [Background] Jeschke MG. The hepatic response to thermal injury: is the liver important for postburn outcomes? Mol Med. 2009 Sep-Oct;15(9-10):337-51. doi: 10.2119/molmed.2009.00005. Epub 2009 Apr 10. PMID 19603107
- [Background] Hew JJ, Parungao RJ, Shi H, Tsai KH, Kim S, Ma D, Malcolm J, Li Z, Maitz PK, Wang Y. Mouse models in burns research: Characterisation of the hypermetabolic response to burn injury. Burns. 2020 May;46(3):663-674. doi: 10.1016/j.burns.2019.09.014. Epub 2019 Oct 10. PMID 31606314
- [Background] Jeschke MG, van Baar ME, Choudhry MA, Chung KK, Gibran NS, Logsetty S. Burn injury. Nat Rev Dis Primers. 2020 Feb 13;6(1):11. doi: 10.1038/s41572-020-0145-5. PMID 32054846
- [Background] Stanojcic M, Abdullahi A, Rehou S, Parousis A, Jeschke MG. Pathophysiological Response to Burn Injury in Adults. Ann Surg. 2018 Mar;267(3):576-584. doi: 10.1097/SLA.0000000000002097. PMID 29408836
- [Background] Yu YM, Tompkins RG, Ryan CM, Young VR. The metabolic basis of the increase of the increase in energy expenditure in severely burned patients. JPEN J Parenter Enteral Nutr. 1999 May-Jun;23(3):160-8. doi: 10.1177/0148607199023003160. PMID 10338224